CLINICAL TRIAL: NCT06430541
Title: Study of Psilocybin Assisted Psychotherapy to Address Fear of Recurrence in Patients Diagnosed With Early-stage Breast Cancer and Ovarian Cancer in Remission
Brief Title: Study of Psilocybin Assisted Psychotherapy to Address Fear of Recurrence
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Usona Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-1455.cc
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Ovarian Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psilocybin Assisted Psychotherapy (Experimental): 25mg cGMP Psilocybin in combination with manualized therapy
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — A tryptamine that produces its behavioral effects primarily by acting as post-synaptic agonists at serotonin 5-HT2A and 5-HT2c receptors.

SUMMARY:
The goal of this clinical trial is to test whether psilocybin along with therapy in women with early breast cancer and ovarian cancer in remission can improve their fear of recurrence. The main question[s] it aims to answer [is/are]:

Does psilocybin assisted therapy improve fear of cancer recurrence? Does psilocybin assisted therapy improve anxiety, depression, and quality of life?

Participants will complete a series of survey measures, participate in preparatory therapy. After prep therapy is complete, they will receive a moderately high dose of psilocybin in a monitored and supportive environment. After the dosing day, they will complete 4 sessions of integrative therapy and complete survey measures.

ELIGIBILITY:
Inclusion Criteria:

1, Aged ≥ 21 2. Diagnosis of:

* early-stage breast cancer at low risk of recurrence

  * defined as clinical stage 1 or 2
  * completed primary treatment (surgery, chemotherapy [adjuvant, patients may continue to be treated with neoadjuvant], and/or radiation) > 6 months ago
  * oncologist reported risk of recurrence at 10 years < 20%
* late-stage ovarian cancer at high risk of recurrence

  * defined as Clinical stage 3 or 4
  * currently in remission
  * oncologist reported risk of recurrence at 10 years > 80% 2. Functional Status defined as:
* Eastern Cooperative Oncology Group (ECOG) ≤1
* Palliative Performance Scale (PPS) ≥60%
* Ability to tolerate PO medication administration 4. Fear of recurrence at screening and baseline 5. Have an identified support person
* Agree to be accompanied home (or to an otherwise safe destination) by the support person, or another responsible party, following dosing 6. Participants of childbearing potential must agree to practice an effective means of birth control throughout the duration of the study.

Exclusion Criteria:

1. Unstable medical conditions or serious abnormalities of complete blood count, chemistries, or EKG that in the opinion of the study physician would preclude safe participation in the trial. Some examples include:

   * Congestive heart failure
   * Valvular heart disease
   * Clinically significant arrhythmias (e.g., ventricular fibrillation, torsades) or clinically significant EKG abnormality (i.e., QTC interval > 450)
   * Recent acute myocardial infarction or evidence of ischemia
   * Malignant hypertension
   * Congenital long QT syndrome
   * Acute renal failure
   * Severe hepatic impairment
   * Respiratory failure
   * eGFR < 50 mL/min/1.73m2
   * LFTs > 1.5 x ULN
   * WBC < 5 x 10*9/L
   * Hemoglobin < 8.0 g/dL
   * Platelets < 150 x 10*9/L
2. Risk for hypertensive crisis defined as:

   Screening and Baseline blood pressure >140/90 mmHg
3. Significant central nervous system (CNS) pathology

   Examples include:
   * Primary or secondary cerebral neoplasm
   * Epilepsy
   * History of stroke
   * Cerebral aneurysm
   * Dementia
   * Delirium
4. Primary psychotic or affective psychotic disorders Examples include current or past DSM-5 criteria for:

   * Schizophrenia spectrum disorders
   * Schizoaffective disorder
   * Bipolar I or bipolar II disorder
   * Major Depressive Disorder with psychotic features
   * Prior history of psychosis due to medical condition or substance use
5. Family history of psychotic or serious bipolar spectrum illnesses.

   Examples include first-degree relative with:
   * Schizophrenia spectrum disorders
   * Schizoaffective disorder
   * Bipolar I disorder with psychotic features
6. High risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation and judgement. Examples include:

   * Agitation
   * Violent behavior
7. Active substance use disorders (SUDs) defined as:

   * DSM-5 criteria for moderate or severe alcohol or drug use disorder (excluding caffeine and nicotine) within the past year
   * DAST-10 score of 3 or higher
   * Two or more "yes" responses to CAGE screening questionnaire
8. Extensive use of serotonergic hallucinogens (e.g., LSD, psilocybin) defined as:

   * Any use in the last 12 months
   * >25 lifetime uses
9. Clinically significant suicidality or high risk of completed suicide defined as:

   * 'Yes' to C-SSRS Suicidal Ideation items 4 or 5 within the last 2 months at Screening or 'since last visit' at Baseline
   * Any C-SSRS Suicidal Behavior item within the past 12 months at Screening or 'since last visit' at Baseline, as defined by 'Yes' to any of the following on the C-SSRS: actual attempt, interrupted attempt, aborted attempt, or preparatory acts
   * Have any suicidal ideation or thoughts, in the opinion of the study physician or PI, that presents a serious risk of suicidal or self-injurious behavior
10. History of hallucinogen persisting perception disorder (HPPD)
11. Pregnancy/lactation
12. Cognitive impairment as defined by:

    • Montreal Cognitive Assessment Test (MoCA) < 23
13. Concurrent Medications

    * Antidepressants
    * Centrally-acting serotonergic agents (e.g., MAO inhibitors)
    * Serotonin-acting dietary supplements (such as 5-hydroxy-tryptophan or St. John's wort)
    * Antipsychotics (e.g., first and second generation)
    * Mood stabilizers (e.g., lithium, valproic acid)
    * Aldehyde dehydrogenase inhibitors (e.g., disulfiram)
    * Significant inhibitors of UGT 1A0 or UGT

      1A10
    * Efavirenz
14. Have a positive urine drug test including Amphetamines, Barbiturates, Buprenorphine, Benzodiazepines, Cocaine, Cannabis, Methamphetamine, MDMA, Methadone, Opiates (Morphine, Oxycodone) unless prescribed, and Phencyclidine (PCP).
15. Have a psychiatric condition judged to be incompatible with establishment of rapport with the study therapists or safe exposure to psilocybin
16. Have any psychological or physical symptom, medication, or other relevant finding , based on the clinical judgment of the PI or relevant clinical study staff that would make a participant unsuitable for the study.
17. Have an allergy or intolerance to any of the materials contained in the drug product
18. Non-English speaking individual
19. Be enrolled in another clinical trial assessing intervention(s) for anxiety, depression, and/or existential distress (e.g., pharmacologic or psychotherapeutic interventions)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Fear of Cancer Recurrence Inventory | 1-week, 4-weeks, 8-weeks* (primary outcome time point), 12-weeks, and 24-weeks.
  Measured by change in core on the Fear of Recurrence Inventory completed at screening and baseline.
  The FCRI's total score ranges from 0 to 36, with higher scores indicating greater FCR severity.

SECONDARY OUTCOMES:
Safety as measured by adverse events | for the duration of study participation -6 months
  Assess Adverse Events, Treatment Emergent Adverse Events, Serious Adverse Events

OTHER OUTCOMES:
Depression | Baseline, 1-week, 4-weeks, 8-weeks, 12-weeks, and 24-weeks
  Symptoms of depression as measured by HADS-D 0-7 (Normal) 8-10 (Mild) 11-15 (Moderate) 16-21 (Severe)
Anxiety | Baseline, 1-week, 4-weeks, 8-weeks, 12-weeks, and 24-weeks
  Symptoms of anxiety as measured by HADS-A 0-7 (Normal) 8-10 (Mild) 11-15 (Moderate) 16-21 (Severe)
Cancer-related Existential Distress | Baseline, 1-week, 4-weeks, 8-weeks, 12-weeks, and 24-weeks
  Demoralization Syndrome will be measured with the Demoralization Scale Version II (DS-II) 16 items that are rated on a three-point Likert scale (0 = never; 1 = sometimes; 2 = often), thus total DS-II scores range from 0-32
Quality of Life-FACT-G | Baseline, 1-week, 4-weeks, 8-weeks, 12-weeks, and 24-weeks
  Quality of life as measured by FACT-G The FACT-G consists of 27 items grouped into four general subdomains: physical well-being (PWB; 7 items, score range: 0-28), social/family well-being (SFWB; 7 items, score range: 0-28), emotional well-being (EWB; 6 items, score range: 0-24), and functional well-being (FWB; 7 items, score range: 0-28).
Spirituality | Baseline, 1-week, 4-weeks, 8-weeks, 12-weeks, and 24-weeks
  Spirituality as measured by FACT-Sp The Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being (FACIT-Sp) scale has a total score range of 0-48. The scale is made up of 12 items, each scored on a 5-point Likert scale with options ranging from 0 ("not at all") to 4 ("very much"). Two items are negatively worded and must be reverse-coded. Higher scores indicate higher well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Fischer, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Outpatient CTRC, Aurora, Colorado
  - University of Colorado Cancer Center, Aurora, Colorado